CLINICAL TRIAL: NCT00971555
Title: Thyroid Function in Late Preterm Infants in Relation to Severity of Illness
Brief Title: Thyroid Function in Late Preterm Infants
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: David A. Paul, MD, Christiana Hospital
Other Study IDs: CCC#29111
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Transient Hypothyroxinemia
Keywords: Transient Hypothyroxinemia; Late Preterm Infants; Total T4; TSH; Illness severity; NICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for total T4 and TSH testing will be done utilizing standardized filter paper used for the State of Delaware Newborn Screening Program.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Late preterm: Late preterm infants admitted to the NICU

SUMMARY:
Transient hypothyroxinemia (TH) is a condition characterized by low levels of serum thyroxine (T4) and normal levels of thyroid stimulating hormone (TSH). TH in premature infants has been found to be related to severity of illness. T4 levels in very low birth weight infants born prematurely has been found to be inversely correlated to severity of illness. In very low birth weight infants, TH has been associated with poor outcomes. Little is known about thyroid function in late preterm infants.

Hypotheses:

1. Ill late preterm infants will have lower total T4 levels than healthy late preterm infants.
2. Total T4 and possibly TSH levels will be inversely correlated with short-term outcomes.
3. Late Preterm infants born by cesarean section will have lower T4 levels compared to those born by vaginal birth.

ELIGIBILITY:
Inclusion Criteria:

* any infant born between 34 0/7 weeks and 36 6/7 weeks gestation born at Christiana Hospital

Exclusion Criteria:

* outborn infants
* infants with major congenital anomalies

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Late preterm infants
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Correlation of total T4 and TSH with gestational age, birth weight, and mode of delivery. | First week of life

CONTACTS AND LOCATIONS:
Overall Officials: Renee M Behme, MD, Principal Investigator — Christiana Hospital; David A Paul, MD, Principal Investigator — Christiana Hospital
Locations (1):
- Christiana Hospital, Newark, Delaware, United States

REFERENCES:
- [Derived] Behme RM, Mackley AB, Bartoshesky L, Paul DA. Thyroid function in late preterm infants in relation to mode of delivery and respiratory support. J Pediatr Endocrinol Metab. 2014 May;27(5-6):425-30. doi: 10.1515/jpem-2013-0243. PMID 24259241